CLINICAL TRIAL: NCT01382563
Title: Registry for Eosinophilic Gastrointestinal Disorders (REGID)
Acronym: EoE
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2010-1579
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Eosinophilic Gastrointestinal Disorders (EGID); Eosinophilic Esophagitis; Eosinophilic Disorder
Keywords: Eosinophilic Gastrointestinal Disorders; EGID; Eosinophilic Esophagitis; Registry; Eosinophils; Eosinophilia; Eosinophilic enteropathy; Eosinophilic enteritis; Eosinophilic gastritis; Eosinophilic gastroenteritis; Eosinophilic gastroenteropathy
MeSH Terms: conditions — Eosinophilic Esophagitis; Eosinophilia; Eosinophilic enteropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Develop Registry tool

DETAILED DESCRIPTION:
The purpose of this research study is to develop a registry tool used for the management and care of patients with eosinophilic disorders, and create a research resource that will provide further insights into these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Eosinophilic Gastrointestinal Disorder diagnosis

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eosinophilic Gastrointestinal Disorders
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Registry Aim | Open-ended
  The registry will allow for the standardization of care while also allowing us to identify gaps in care that need to be addressed and areas for future research at Cincinnati Children's Hospital Medical Center (CCHMC) and collaborating sites around the nation.

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (8):
- United States (8):
  - Rady Children's Hospital, San Diego, California
  - The Children's Hospital, Aurora, Colorado
  - Northwestern University School of Medicine, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - University of North Carolina, Chapel Hill, North Carolina
  - Kara Kliewer, Mason, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- See also: Registry for Eosinophilic Gastrointestinal Disorders — https://www.regid.org/